CLINICAL TRIAL: NCT00899561
Title: Correlation Between Middle Turbinate Histopathology and Computed Tomography Staging in Chronic Rhinosinusitis
Brief Title: Computed Tomography (CT) Score and Histopathology of the Middle Turbinate in Chronic Rhinosinusitis
Acronym: CT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: MeirMc
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Rhinosinusitis
Keywords: Chronic rhinosinusitis; Computed tomography; Histology; Middle turbinate; Morphometry; osteomyelitis; polyps
MeSH Terms: conditions — Osteomyelitis; Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Middle turbinate samples of patients with limited, intermediate, and extensive chronic sinus disease.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In a previous study (Berger el al. Old and new aspects of middle turbinate histopathology. Otolaryngol Head Neck Surg. 2009;140:48-54), the investigators reported significant histopathologic changes in the middle turbinate mucosa of patients with chronic rhinosinusitis compared with normal controls. However, patients' mean Lund-MacKay CT score was 6.5±6.7 and were considered as having a relatively limited sinus disease (a score of 1-8). Nine to sixteen was considered as intermediate sinus disease, and 17-24 extensive. No osteomyelitic changes were seen in this study group.

The investigators hypothesize that a comparison between the three groups of patients with chronic rhinosinusitis having limited, intermediate, and extensive sinus disease would show that the higher the CT staging, the greater the histopathologic changes of the middle turbinate. The investigators also expect to find osteomyelitic changes in the middle turbinate of patients with higher CT staging.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with chronic rhinosinusitis who failed conservative medical treatment,
* Patients who stopped treatment (topical or systemic corticosteroids) at least two months before endoscopic sinus surgery.

Exclusion Criteria:

* Immunosuppressed patients,
* Patients in whom no indication to excise the middle turbinate was found, AND
* Patients in whom a pathologic evaluation of the middle turbinate was necessary (e.g., suspected neoplastic disorder).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a limited (of 1-8), intermediate (9-16), and extensive (17-24) sinus disease.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
inflammation of soft tissue and bony elements of the middle turbinate | two years

SECONDARY OUTCOMES:
correlation between middle turbinate histopathology and CT staging in chronic rhinosinusitis | two years

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Berger, MD, Principal Investigator — Meir Medical Center; Roee Landsberg, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel